CLINICAL TRIAL: NCT00067314
Title: A Phase II Study Of Intravenous Edotecarin (PHA-782615) In Patients With Anthracycline- And Taxane Resistant Metastatic Breast Cancer
Brief Title: Study in Women With Metastatic Breast Cancer Whose Cancer Has Gotten Worse After Anthracycline and Taxane Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDOABC-4439-001
Record Dates: First submitted 2003-08-15; First posted 2003-08-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — edotecarin

INTERVENTIONS:
Drug: Edotecarin

SUMMARY:
This international study will study how metastatic breast cancer responds to the investigational drug treatment, what are the side effects of the investigational drug when given to women with metastatic breast cancer and how often do these side effects occur. The study will also analyze how fast investigational drug and its breakdown products are cleared from the blood in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic breast cancer not amenable to surgery or radiation with curative intent
* Must have received any chemotherapy regimen in the past
* Evidence of tumor resistance to last chemotherapy defined as progression after 6 months of previous chemotherapy for advanced disease
* Must have measurable (by imaging techniques) disease
* Adequate bone marrow, liver and renal function
* Must provide evidence of informed consent and willingness and ability to comply with scheduled visits, treatment plan and study procedures.

Exclusion Criteria:

* Received more than 2 prior chemotherapy regimens for metastatic disease
* Received in the past another drug of the same class as the investigational drug, i.e. topoisomerase I inhibitor
* Enrolled in another clinical intervention study
* Pregnancy, breast feeding, fertile women refusing to use reliable contraceptive methods
* Cardiac or thrombotic event in the last 12 months
* Brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor activity of single-agent Edotecarin by determining the objective response rate

SECONDARY OUTCOMES:
Time to tumor response (TAR)
Duration of response (DR)
Time to tumor progression (TTP)
Time to treatment failure (TTF)
Overall survival (OS)
Clinical benefit
ie, a composite profile of pain intensity
analgesic consumption and performance status (pain and analgesic consumption to be measured as described in Purohit 1994 [18]
performance status to be assessed using the Eastern Cooperative Oncology Group ([ECOG]) scale [Appendix 2]
Overall safety profile characterized by type, frequency, severity (as graded by version 2.0 of the National Cancer Institute (NCI) Common Toxicity Criteria [CTC]
[Appendix 3], timing and relationship to study therapy of adverse events and laboratory abnormalities.
Plasma pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (6):
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Orange, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Nashville, Tennessee
- Australia (2):
  - Pfizer Investigational Site, East Bentleigh, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Haine-Saint-Paul
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Wilrijk
- France (5):
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EDOABC-4439-001&StudyName=Study%20in%20Women%20with%20Metastatic%20Breast%20Cancer%20whose%20Cancer%20has%20Gotten%20Worse%20after%20Anthracycline%20and%20Taxane%20Therapy